CLINICAL TRIAL: NCT05291403
Title: The Efficacy and Safety Study of Medical Thoracoscope Cryotherapy Combined With Standard First-line Treatment of Advanced Non-small Cell Lung Cancer and Malignant Pleural Effusion: a Multicenter, Prospective, Randomized, Controlled Clinical Trial
Brief Title: Efficacy and Safety Study of Medical Thoracoscope Cryotherapy Combined Standard First-line Treatment of Advanced Non-small Cell Lung Cancer and Malignant Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qian Qi, Doctor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2-21-QFS
Record Dates: First submitted 2022-02-22; First posted 2022-03-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: advanced Non-small Cell Lung Cancer; Malignant Pleural Effusion; Thoracoscopy; Cryotherapy Effect
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (medical thoracoscopic cryotherapy) (Experimental)
  Interventions: Other: Medical thoracoscopic cryotherapy combined with standard first-line therapy for advanced non-cell lung cancer
- Cisplatin/erythromycin control group (sequential intrathoracic injection of cisplatin/erythromycin) (Active Comparator)
  Interventions: Other: Sequential intrathoracic injection of cisplatin/erythromycin combined with standard first-line therapy for advanced non-cell lung cancer
- Blank control group (Other): Only intrathoracic tube was used to drain pleural effusion, and local pleural cavity was not treated.
  Interventions: Other: Standard first-line therapy for advanced non-cell lung cancer without intrathoracic treatment

INTERVENTIONS:
Other: Medical thoracoscopic cryotherapy combined with standard first-line therapy for advanced non-cell lung cancer — Medical thoracoscopic cryotherapy: medical thoracoscopy biopsy hole insert bendable freezing probes, place the frozen probe placed in the center of the tumor at the top will be frozen carbon dioxide gas source pressure adjustment to the bar of 50-60 bar, tread down switch, foot pedal to start the probe, after about 30 s at the top of the probe to form a ice hockey, local tissue after frozen white, sometimes a small amount of bleeding; Fix the probe, loosen the pedal, and wait 30 seconds for automatic melting and rewarming (bleeding probability is low after full rewarming). Freeze 5 to 10 at a time.
  In addition, all patients were treated with standard first-line regimens according to guidelines of non small cell lung cancer (NSCLC) and Eastern Cooperative Oncology Group (ECOG) scores.
  Arms: Experimental group (medical thoracoscopic cryotherapy)
Other: Sequential intrathoracic injection of cisplatin/erythromycin combined with standard first-line therapy for advanced non-cell lung cancer — The pleural effusion was fully drained and cisplatin 40mg/m2 was given, dissolved in 100mL 0.9% sodium chloride (NaCl) solution 100 mL, then injected into the pleural cavity and retained for 24 hours. Erythromycin was sequentially injected into the thorax to seal the pleural cavity.
  In addition, all patients were treated with standard first-line regimens according to guidelines of NSCLC and ECOG scores.
  Arms: Cisplatin/erythromycin control group (sequential intrathoracic injection of cisplatin/erythromycin)
Other: Standard first-line therapy for advanced non-cell lung cancer without intrathoracic treatment — Only intrathoracic tube was used to drain pleural effusion, and local pleural cavity was not treated.
  In addition, all patients were treated with standard first-line regimens according to guidelines of NSCLC and ECOG scores.
  Arms: Blank control group

SUMMARY:
This study intends to investigate the efficacy and safety of medical thoracoscopic cryotherapy combined with standard first-line treatment of advanced non-small cell lung cancer with malignant pleural effusion through a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. Non-small cell lung cancer with pleural metastasis confirmed by histopathology or cytology;
3. ECOG score 0-1;
4. Cardiopulmonary function can tolerate painless thoracoscopic examination;
5. Patients who underwent medical thoracoscopy for pleural effusion at first diagnosis and underwent medical thoracoscopy cryotherapy at the same time of biopsy were also included in the study. Non-small cell lung cancer was confirmed by pathological results;
6. All subjects or their guardians must sign the informed consent before entering the study.

Exclusion Criteria:

1. Expected survival <2 months;
2. Hemoglobin <110g/L, white blood cell count <3×109/L, neutrophil <2.0×109/L, platelet <100×109/L;
3. severe cardiac insufficiency, abnormal liver and kidney function (blood test results of transaminase and creatinine > 1.5 times the normal upper limit);
4. have received chemotherapy or anti-angiogenic drugs (such as bevacizumab, endu, anlotinib, etc.);
5. History of radiotherapy;
6. history of intrathoracic local treatment;
7. multiple serous cavity effusion, or bilateral pleural effusion;
8. patients allergic to erythromycin;
9. the lung cannot be reopened.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pleural progression free survival, P-PFS | up to 2 months
  According to Millar's criteria, P-PFS was defined as absence of pleural effusion lasting more than 4 weeks; Or an order of magnitude reduction in pleural effusion (such as large to medium volume, or medium to small volume) lasting more than 4 weeks; Or pleural effusion with no significant change, lasting more than 4 weeks.

SECONDARY OUTCOMES:
Total effective rate | up tp 2 months
  Complete remission (CR) : pleural effusion disappeared and lasted for more than 4 weeks; Partial remission (PR) : reduction of pleural effusion by 1 order of magnitude (e.g., large to medium volume, or medium to small volume) for more than 4 weeks; CR+PR was denoted as the total effective rate.
Progression-free survival (PFS) | up to 2 months
modified Medical Research Council Dyspnea Scale | up to 2 months
  The modified Medical Research Council Dyspnea Scale (mMRC) is used to assess degree of baseline functional disability due to dyspnea. The minimum and maximum values are 0 and 4, and higher scores mean a worse outcome. Score 0 means dyspnea only with strenuous exercise; score 1 means dyspnea when hurrying or walking up a slight hill; score 2 means walks slower than people of the same age because of dyspnea or has to stop for breath when walking at own pace; score 3 means stops for breath after walking 100 yards (91 m) or after a few minutes; score 4 means too dyspneic to leave house or breathless when dressing.
Overall survival time | up to 2 months
Adverse reactions | up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory, The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No